CLINICAL TRIAL: NCT04054271
Title: Effects of ABO Blood Types on the Survival and Marginal Bone Resorption of Dental Implants
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, PhD, DDA, Assistant professor, Yuzuncu Yil University
Other Study IDs: 29112017/05
Record Dates: First submitted 2019-08-06; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Implant Tissue Failure
Keywords: Blood types, Dental implant, Marginal Bone Resorption, Implant Survival

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates implant survival and marginal bone resorption in patients receiving implant treatment with respect to demographic data and AB0 (groups) blood types.

DETAILED DESCRIPTION:
For a successful dental implant, optimal soft and hard tissue characteristics are required. These characteristics include appropriate bone quality and a healthy adherent keratinized gingiva that surrounds the implant neck. The most common complications are peri-implant diseases and marginal bone loss for dental implants. Marginal bone loss around the implant may be observed as a long-term complication due to microbial dental plaque-induced peri-implant inflammatory disease or may be observed in the absence of such a disease.

The immune system and genetic factors are known to have important effects on implant success, and ABO blood types are also included in the genetic factors. In the studies evaluating the association of ABO blood types with increased susceptibility to infection and various systemic diseases, it was reported that the percentages of blood types differed significantly, especially in skeletal-muscle system injuries, fractures and cardiovascular disease susceptibility. Also some researchers reported that blood types may be effective on the bacteria colonization which is the main reason of the periodontal diseases. ABO blood types may have an impact on dental implant success and survival.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study group included being 18 years of age and non-smoker, not having any systemic disease, not having undergone any hard and soft tissue augmentation during implant surgery, having implants placed at bone level, having received cylindrical form implants with SLA surface structure, not missing any follow-up visits after implant surgery evidenced with radiographic recordings, having received flat abutment, having cemented implants, and being rehabilitated with fixed prosthetic restoration.

Exclusion Criteria:

* No

Ages: 19 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study was performed on patients who had undergone implant treatment and had prosthetic rehabilitation at the Faculty of Dentistry of the Van Yuzuncu Yil University between 2010 and 2017 and who had been followed up for at least one year.
Sampling Method: Non-Probability Sample
Enrollment: 963 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Marginal bone resorption measurements (mm) in dental implants. | 1 year
  We evaluated marginal bone resorption in patients receiving implant treatment with respect to ABO blood types. These measurements will be measured by periapical radiographs. Periapical radiographs were taken with a parallel technique to measure the amount of mesial and distal bone resorption in the neck region of the implants.
Implant survival rates according to demographic data | 1 year
  We evaluated implant survival rates by age and sex on a yearly basis

CONTACTS AND LOCATIONS:
Locations (1):
- Serap Keskin Tunc, Van, Turkey (Türkiye)